CLINICAL TRIAL: NCT04742101
Title: Phase I / II, Open Label, Dose Escalation Part (Phase I) Followed by Non-comparative Expansion Part (Phase II), Multi-centre Study, Evaluating Safety, Pharmacokinetics and Efficacy of S65487, a Bcl2 Inhibitor Combined With Azacitidine in Adult Patients With Previously Untreated Acute Myeloid Leukemia Not Eligible for Intensive Treatment
Brief Title: Phase I/II Trial of S65487 Plus Azacitidine in Acute Myeloid Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut de Recherches Internationales Servier (Other)
Collaborators: ADIR, a Servier Group company (Industry)
Responsible Party: Sponsor
Organization: Servier (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL1-65487-003; 2020-003061-19 (EudraCT Number)
Record Dates: First submitted 2020-12-14; First posted 2021-02-05 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; Dose escalation; Phase I/II; Azacitidine; Combination; Oncology
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Neoplasms | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- S65487 with azacitidine (Experimental)
  Interventions: Drug: S65487 and azacitidine

INTERVENTIONS:
Drug: S65487 and azacitidine — Treatment cycle of combination of S65487 and azacitidine during 4 weeks. Two administration schedules are set up. S65487 will be administered via intravenous (IV) infusion. Azacitidine will be administered via either subcutaneous (SC) or Intravenous (IV) infusion according to local practices.

SUMMARY:
The purpose of this study is to assess the safety, tolerability and clinical activity of the combination S65487 with azacitidine in patients with acute myeloid leukaemia.

DETAILED DESCRIPTION:
The study is designed in two parts: A dose escalation phase I part, and a dose expansion phase II part with an additional potential expansion cohort.

During dose escalation of S65487 in combination with azacitidine, only S65487 agent dose will escalate and a DDI (Drug-Drug interaction) assessment between S65487 and posaconazole (antifungal drug) will be performed. A ramp-up dose of S65487 will be administered on the first two days of cycle 1, then the full dose of S65487 will be administered for the remainder of cycle 1. Each treatment cycle is 28 days.

For the expansion phase, the dose will be the RP2D (Recommended Phase 2 Dose) determined during phase I part. An additional potential expansion cohort will be included if there is more than one promising dose/schedule candidate.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participant aged ≥ 18 years old
* Participants with cytologically confirmed and documented treatment naïve, de novo or secondary AML defined by WHO 2016 classification (Arber, 2016). Secondary AML includes:

  * Previous myelodysplastic syndrome transformed
  * AML due to exposure to potentially leukemogenic therapies or agents (e.g. radiation therapy, alkylating agents, topoisomerase II inhibitors) with the primary malignancy in remission for at least 3 years
* Participants not eligible for standard induction chemotherapy

  * Aged ≥ 75 years old
  * Or Age ≥18 years with at least one of the following comorbidities:

    * Clinically significant heart or lung comorbidities, as reflected by at least one of:

      * Lung diffusing capacity for carbon monoxide (DLCO) ≤65% of expected
      * Forced expiratory volume in 1 second (FEV1) ≤65% of expected
    * Other contraindication(s) to anthracycline therapy (must be documented)
    * Other comorbidity that the Investigator judges as incompatible with intensive remission induction chemotherapy, which must be documented
* ECOG (Eastern Cooperative Oncology Group) performance status should be (criterion should be rechecked at inclusion visit) ECOG ≤ 2.
* Written informed consent obtained prior any study-specific procedure as described in section 13.3 of the protocol.
* Adequate renal and hepatic function
* Circulating White Blood Cell Count (WBC count) < 25*109 G/L (with or without use of hydroxycarbamide/leukapheresis)
* Serum potassium, serum calcium, serum phosphates, serum magnesium within normal limits with or without supplementation.

Exclusion Criteria:

* Major surgery within 3 weeks prior to the first IMP administration, or participants who have not recovered from side effects of the surgery
* Any radiotherapy within 3 weeks before the first IMP administration,
* Allogenic stem cell transplant within 3 months before the first IMP administration and/or participants with active Graft-versus-host disease within 3 months before the first IMP administration and/or participants who still receive immunosuppressive treatment within 3 months before the first IMP administration and/or participant who receive donor lymphocyte infusion (DLI) within 3 months before the first IMP administration
* Acute promyelocytic leukemia (APL, French-American-British M3 classification)
* Favorable risk cytogenetics such as t(8;21), inv(16) or t(16;16) or t(15;17) as per the National Comprehensive Cancer Network (NCCN) Guidelines Version 3, 2019 for Acute Myeloid Leukemia
* Treatment with hypomethylating agents (decitabine/azacitidine) or Venetoclax for AHD (antecedent hematologic disorders) in the 3 months prior to the first IMP intake

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) (phase I part) | Through the end of first cycle (each cycle is 28 days)
  DLT assessment at the end of cycle 1
Adverse Event (phase I part) | Through study completion, an average of 3 years ans 5 months
  AE recording throughout the study evaluated according to CTCAE v5.0, dose interruptions, reductions, and intensity
Complete Remission (CR) rate (phase II part) | Through study completion, up to 3 years and 5 months
  CR rate is defined as the proportion of subjects who achieve complete response. Response is evaluated based on the "'Diagnosis and management of AML in adults: 2022 ELN recommendations from an international expert panel" (Döhner, 2022).

SECONDARY OUTCOMES:
PharmacoKinetics - maximum Concentration at the End of the infusion (Cinf) (phase I and phase II parts) | Cycle 1 Day 1, Cycle 1 Day 8, Cycle 1 Day 15 (schedule 1, first two cohorts), Cycle 2 Day 8 (from Cohort 3), or Day 15 (first two cohorts)(each cycle is 28 days)
  PK parameters of S65487, azacitidine and potential metabolite(s)
PharmacoKinetics - Area Under the Curve (AUC) (phase I and phase II parts) | Cycle 1 Day 8 to Day 9, Cycle 2 Day 8 to Day 9 (from cohort 3), or Day 15 to Day 16 (first two cohorts)(each cycle is 28 days)
  PK parameters of S65487, azacitidine and potential metabolite(s)
Assessment of anti-leukemic activity of S65487 combined to azacitidine (phase I and phase II parts) | Through study completion, an average of 3 years and 5 months
  Complete Remission rate
Assessment of anti-leukemic activity of S65487 combined to azacitidine (phase I and phase II parts) | Through study completion, an average of 3 years and 5 months
  Progression Free Survival

CONTACTS AND LOCATIONS:
Locations (11):
- Institut Gustave Roussy, Villejuif, France
- Semmelweis Egyetem Belgyógyászati és Onkológiai Klinika Klinikai Farmakológiai Részleg, Budapest, Hungary
- Narodowy Instytut Onkologii im. M. Sklodowskiej-Curie Klinika Transplantacji Szpiku i Onkohematologii pokoj 4.041 ul. Wybrzeze Armii Krajowej 15, Gliwice, Poland
- South Korea (2):
  - Seoul National University Hospital - Department of Hematology-Oncology, Seoul
  - Samsung Medical Center - Division of Hematology-Oncology, Seoul
- Spain (3):
  - Hospital 12 de Octubre Servicio de Hematología, Madrid
  - C. Universidad de Navarra Servicio de Hematologia, Pamplona
  - H. Universitario La Fe Servicio de Hematologia, Valencia
- United Kingdom (3):
  - Western General Hospital, Edinburgh
  - University College London - Hospitals NHS Foundation Trust, London
  - The Christie NHS foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Qualified scientific and medical researchers can request access to anonymized patient-level and study-level clinical trial data.
  Access can be requested for all interventional clinical studies:
  * used for Marketing Authorization (MA) of medicines and new indications approved after 1 January 2014 in the European Economic Area (EEA) or the United States (US).
  * where Servier is the Marketing Authorization Holder (MAH). The date of the first MA of the new medicine (or the new indication) in one of the EEA Member States will be considered for this scope.
  In addition, access can be requested for all interventional clinical studies in patients:
  * sponsored by Servier
  * with a first patient enrolled as of 1 January 2004 onwards
  * for New Chemical Entity or New Biological Entity (new pharmaceutical form excluded) for which development has been terminated before any Marketing authorization (MA) approval.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After Marketing Authorisation in EEA or US if the study is used for the approval.
Access Criteria: Researchers should register on Servier Data Portal and fill in the research proposal form. This form in four parts should be fully documented. The Research Proposal Form will not be reviewed until all mandatory fields are completed.
URL: https://clinicaltrials.servier.com/

REFERENCES:
- [Background] Pierola AA, De Botton S, Jan JH, Campbell V, O'Nions J, Calbacho M, Ervin-Hayes AL, Keagle K, Maillard A, Beneton M, Romagnoli M, Broniscer A. Trial in Progress: An Open Label Phase I/II, Multicenter Study Evaluating Safety, Pharmacokinetics and Efficacy of S65487, a BCL-2 Inhibitor Combined with Azacitidine in Adults with Previously Untreated Acute Myeloid Leukemia Ineligible for Intensive Treatment. Blood. 2023 Nov 2;142(Supplement 1):1555. doi: https://doi.org/10.1182/blood-2023-180795
- See also: Find Results on Servier Clinical Trial Data website — https://clinicaltrials.servier.com/
- Available data/document: Individual Participant Data Set — https://clinicaltrials.servier.com/
- Available data/document: Study Protocol — https://clinicaltrials.servier.com/
- Available data/document: Statistical Analysis Plan — https://clinicaltrials.servier.com/
- Available data/document: Informed Consent Form — https://clinicaltrials.servier.com/
- Available data/document: Clinical Study Report — https://clinicaltrials.servier.com/
- Available data/document: Study-level clinical trial data — https://clinicaltrials.servier.com/